CLINICAL TRIAL: NCT02818972
Title: A Prospective, Multicenter, Non-Blinded, Non-Randomized Study of the RelayPro Thoracic Stent-Graft in Subjects With Thoracic Aortic Aneurysms and Penetrating Atherosclerotic Ulcers
Brief Title: RelayPro Thoracic Stent-Graft in Subjects With Thoracic Aortic Aneurysms and Penetrating Atherosclerotic Ulcers
Acronym: RelayPro-A
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bolton Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-0015-16
Record Dates: First submitted 2016-06-27; First posted 2016-06-30 (Estimated); Last update posted 2025-05-31 (Actual); Status verified 2025-04

CONDITIONS: Aortic Aneurysm, Thoracic; Penetrating Ulcer
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Penetrating Atherosclerotic Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- RelayPro (Experimental): Endovascular treatment with the investigational device.
  Interventions: Device: RelayPro

INTERVENTIONS:
Device: RelayPro — Endovascular treatment with investigational device.

SUMMARY:
Investigate the safety and effectiveness of the RelayPro Thoracic Stent-Grafts in subjects with thoracic aortic aneurysms (TAA) and penetrating atherosclerotic ulcers (PAU) of the descending thoracic aorta.

DETAILED DESCRIPTION:
The objective of this study is to investigate the safety and effectiveness of the RelayPro Thoracic Stent-Grafts in subjects with thoracic aortic aneurysms and penetrating atherosclerotic ulcers of the descending thoracic aorta.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 18 years of age
* Subject has specified disease in his/her descending thoracic aorta.
* Subject have anatomical compliance for the device specified for both access vessels and treatment area.
* Subject must be willing to comply with the follow-up evaluation schedule.
* Subject (or Legally Authorized Representative) agrees an Informed Consent Form prior to treatment.

Exclusion Criteria:

* Subject has specified disease of the thoracic aorta which is not included in the trial, for example: aortic dissection, intramural hematoma, traumatic injury or transection, aortic false aneurysm, ruptured aneurysm.
* Subject anatomy with significant stenosis, calcification, thrombus or tortuosity.
* Subjects with specified compromised circulation.
* Subjects with specified prior procedures.
* Subjects with allergy to contrast media or device components.
* Subjects with disease, for example: suspected connective tissue disorder, specified coagulation disorders, specified coronary artery disease, severe congestive heart failure, stroke and/or Myocardial Infarction (MI) as specified, specified pulmonary disease, specified renal failure.
* Subjects that are pregnant or planning to become pregnant during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Major Adverse Events (MAEs) | 30 days
  Primary safety endpoint is a composite of the following MAEs occurring through 30 days:
  * Death
  * Stroke (excluding transient ischemic attack)
  * Paralysis (excludes paraparesis)
Technical success | 24 hours
  Primary effectiveness rate as measured by the technical success through 24 hours, defined as:
  * Successful delivery of the device through the vasculature;
  * Successful deployment of the device at the intended location; Absence of Type I or III endoleaks; Patent stent-graft without significant stenosis.
Stent graft patency | 12 months
  Primary effectiveness as measured by the rate of stent-graft patency through 12 months.
Aneurysm rupture | 12 months
  Primary effectiveness as measured by the absence of aneurysm rupture through 12 months.
Absence of Type I and III endoleak through 12 months; | 12 months
  Primary effectiveness as measured by the absence of Type I and III endoleak through 12 months.
Absence of stent fractures in the attachment zone through 12 months | 12 months
  Primary effectiveness as measured by the absence of stent fractures in the attachment zone through 12 months.
Absence of open or endovascular secondary interventions | 12 months
  Primary effectiveness as measured by the absence of open or endovascular secondary interventions related to the device or treated pathology through 12 months.
Absence of aneurysm expansion (> 5 mm diameter increase) | 12 months
  Primary effectiveness as measured by the absence of aneurysm expansion (> 5 mm diameter increase) through 12 months, compared to the first post-procedural computed tomographic (CT) imaging study.
Absence of stent-graft migration | 12 months
  Primary effectiveness as measured by the absence of stent-graft migration (> 10 mm) through 12 months, compared to the first post-procedural CT.

SECONDARY OUTCOMES:
Loss of stent-graft patency | 1 month and 6 months
  Loss of stent-graft patency will be assessed with CT scans, or MRIs for subjects unable to tolerate contrast media.
Rate of aneurysm rupture | 1 month and 6 months
  The rate of aneurysm rupture through 1 month and 6 months will be assessed by review of CT or MRI imaging, in addition to site reported adverse events.
Rate of endoleaks of all types | 1 month, 6 months and 12 months
  Persistence of blood flow outside the lumen of the stent-graft but within the native aorta or adjacent vascular segment being treated by the stent-graft will be assessed by CT scans or MRIs for subjects unable to tolerate contrast media.
Rate of stent fractures in the attachment zone | 1 month and 6 months
  Stent fractures in the attachment zone will be assessed at each follow-up visit with CT scans, or MRIs for subjects unable to tolerate contrast media.
Incidence of open or endovascular secondary interventions | 1 month and 6 months
  Secondary effectiveness will be measured by the incidence of open or endovascular secondary interventions related to the device or treated pathology (ie, interventions to treat malperfusion, rupture, aneurysm formation, or aortic expansion).
Rate of aneurysm expansion | 1 month and 6 months
  The rate of aneurysm expansion (> 5 mm diameter increase) assessed by comparison of follow-up imaging to the first post-procedural CT
Rate of stent-graft migration | 1 month and 6 months
  The rate of stent-graft migration (> 10 mm) assessed by comparison of follow-up imaging to the first post-procedural CT.
Individual outcomes of composite MAEs | 6 months and 12 months
  Secondary effectiveness as measured by the individual outcomes of the composite safety endpoints (death, stroke, paralysis), as well as myocardial infarction (MI), renal failure, respiratory failure, bowel ischemia, and procedural blood loss >1,000 cc.
Rate of vascular access complications | During the initial implant attempt
  Secondary effectiveness as measured by the rate of vascular access complications reported during the Treatment visit (stent-graft implant). Outcome measures include successful delivery and deployment of the device, as well as withdrawal of the delivery system.
Duration of implant procedure | Treatment Visit
  Duration of the initial implant procedure captured as the number of minutes from introduction of device to removal of delivery system.
Number of blood transfusions | Treatment Visit through Discharge Visit
  Number of transfusions (units) required from the time of implant through hospital discharge.
Duration of hospitalization | Treatment Visit through Discharge Visit
  Length of hospital stay defined as number of days subject was hospitalized for the initial implant procedure.
Time in Intensive Care Unit (ICU) | Treatment Visit through Discharge Visit
  Duration of time in hours that subject was admitted to the Intensive Care Unit (ICU) following the implant procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Szeto, MD, Principal Investigator — Penn Presbyterian; Venkatesh Ramaiah, MD, Principal Investigator — Arizona Heart Institute
Locations (35):
- United States (24):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Arizona Heart Institute, Phoenix, Arizona
  - University of California, Irvine, Irvine, California
  - Long Beach Memorial Hospital, Long Beach, California
  - Hartford Hospital, Hartford, Connecticut
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University Health, Indianapolis, Indiana
  - St. Vincent Heart Center, Indianapolis, Indiana
  - University of Iowa Hospital and Clinic, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center / Harvard Medical School, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University Hospitals, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania Medical Center / Penn Presbyterian, Philadelphia, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Centennial Heart & Vascular Institute Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Baylor Scott & White Medical Center - Plano The Heart Hospital, Plano, Texas
  - Baylor Scot & White Medical Center - Temple, Temple, Texas
- Japan (11):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Teine Keihinkai Hospital, Sapporo, Hokkaido
  - Nara Medical University Hospital, Kashihara, Nara
  - Niigata University Medical & Dental Hospital, Niigata, Niigata
  - Oita University Hospital, Yufu, Oita Prefecture
  - Morinomiya Hospital, Joto-ku, Osaka
  - National Cerebral & Cardiovascular Center, Suita, Osaka
  - Jichi Medical University Saitama Medical Center, Ōmiya, Saitama
  - Jikei University Hospital, Minato-Ku, Tokyo
  - Keio University Hospital, Shinjuku-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Szeto WY, Vallabhajosyula P, Matsuda H, Moainie SL, Sharafuddin MJ, Corvera J, Smolock CJ, Miyamoto S, Naslund T, Ramaiah V; RelayPro-A Investigators. One-year results with a low-profile endograft in subjects with thoracic aortic aneurysm and ulcer pathologies. J Thorac Cardiovasc Surg. 2022 May;163(5):1739-1750.e4. doi: 10.1016/j.jtcvs.2021.10.071. Epub 2022 Feb 1. PMID 35241276